CLINICAL TRIAL: NCT05996159
Title: Pulmonary Vein Isolation Strategy of Very High Power Short Duration in Patients With Paroxysmal Atrial Fibrillation: Q-INDEX Trial
Brief Title: Pulmonary Vein Isolation Strategy of Very High Power Short Duration in Patients With Paroxysmal Atrial Fibrillation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Q-INDEX
Record Dates: First submitted 2023-08-01; First posted 2023-08-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- vHPSD ablation only for PVI (Experimental): Pulmonary vein encirclement is achieved using contiguous applications of very high power and short duration (90 W over 4 seconds). The inter-lesion distance is set at 3-4mm for the roofs and anterior segments, and 5-6mm for other segments. If the esophageal temperature rises > 38 for segments near the esophagus, encirclement will be applied at 25 W for 15 seconds.
  Interventions: Device: QDOT MicroTM catheter
- vHPSD and AI-guided ablation for PVI (Experimental): At the anterior segments, pulmonary vein encirclement is achieved through contiguous applications using AI-guided ablation (40-50 W, AI target 500, and an inter-lesion distance of 4mm).
  In the other segments, pulmonary vein encirclement is achieved through contiguous applications using very high-power and short-duration techniques (90 W over 4 seconds, inter-lesion distance of 3-4mm; if the segments are near the esophagus, encirclement will be applied at 25 W for 15 seconds).
  Interventions: Device: QDOT MicroTM catheter; Device: AI-guided ablation only for PVI
- AI-guided ablation only for PVI (Experimental): Pulmonary vein encirclement is achieved through contiguous applications using AI-guided ablation (40-50 W, AI target 500 for anterior segments and 400 for other segments, with an inter-lesion distance of 4mm; if the segments are near the esophagus, encirclement will be applied at 25 W for 15 seconds)
  Interventions: Device: AI-guided ablation only for PVI

INTERVENTIONS:
Device: QDOT MicroTM catheter — Novel high power-short duration ablation catheter for atrial fibrillation
  Arms: vHPSD ablation only for PVI; vHPSD and AI-guided ablation for PVI
Device: AI-guided ablation only for PVI — Ablation is the removal or destruction of something from an object by vaporization, chipping, erosive processes, or by other means.
  Arms: AI-guided ablation only for PVI; vHPSD and AI-guided ablation for PVI

SUMMARY:
This study aims to investigate the effect of reducing ablation time for a hybrid approach of vHPSD and AI-guided ablation using the QDOT Micro catheter in PVI among patients with PAF.

DETAILED DESCRIPTION:
Radiofrequency catheter ablation has become a cornerstone strategy for the rhythm control of AF. During the last decade, catheter technology has revolutionized and, accordingly, clinical outcomes after the ablation and procedural efficacy have been improved.

In recent years, the use of the CLOSE protocol employing contiguous, closely spaced applications and targeted ablation index (AI) values has translated into robust acute and long-term success rates for PVI, typically with the power delivery of up to 35 W, and more recently with 40 to 50 W, in power and temperature-controlled mode.

Contiguous ablation using very high-power, short-duration ablation at 90 W over 4 seconds is expected to shorten procedure time. However, changes in lesion geometry and the altered impact of catheter stability on lesion quality may influence procedural efficiency, safety, and effectiveness.

The Q-FFICIENCY trial showed that the vHPSD (90 W, 4 sec), temperature-controlled radiofrequency ablation (25/50 W) has comparable efficacy to conventional-power temperature-controlled ablation.

However, the efficacy of vHPSD ablation may depend on PV thickness due to its lesion characteristics. Therefore, AI-guided ablation may have merits over vHPSD ablation in thickened PV segments. According to the POWER PLUS trial, the proportion of 1st-pass PVI with vHPSD ablation was numerically lower than that of the conventional ablation, although there was marginal significance; 83.9% vs. 90.0%, p-value =0.085.

According to the OPTIMUM trial, a study conducted by our group, roof and anterior walls of the left atrium often require higher AI targets due to their thickness.

Therefore, a hybrid approach that combines both vHPSD and AI-guided ablations according to PV segments may achieve both high efficacy and short ablation time for PVI. The investigators of the POWER PLUS trial also speculated that the hybrid approach based on tissue thickness might offer the optimal balance of procedural efficacy.

However, up to date, no studies have investigated the efficacy and safety of the hybrid approach for PVI. More data is needed to suggest that the hybrid approach could be useful for PVI.

Therefore, this study aims to investigate the effect of reducing ablation time for a hybrid approach of vHPSD and AI-guided ablation using the QDOT Micro catheter in PVI among patients with PAF.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing PVI for PAF

Exclusion Criteria:

* Aged less than 19 years
* Patients with persistent AF
* Patients with previous ablation or surgery for AF
* Patients with intracardiac thrombus or thromboembolic events within the previous 90 days
* Patients with cardiac surgery or acute coronary syndrome within the previous 90 days
* Patients with contraindication(s) for using oral anticoagulants
* Patients with LA anteroposterior diameter of more than 55 mm
* Patients with left ventricular ejection fraction less than 35%
* Pregnants or those who plan to become pregnant during the study
* Life expectancy less than a year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Time for AF ablation | up to 12 months
  Including total PVI time, total ablation time, fluoroscopic time, and total procedure time.

SECONDARY OUTCOMES:
Acute PV reconnection rate | up to 12 months
  Including residual PV potential and early reconnection after 1st pass PVI.
The segment of residual PV potential | up to 12 months
  Descript as RSPV roof/anterior/posterior/carina, RIPV anterior/posterior/inferior/carina, LSPV roof/anterior(ridge)/posterior/carina, LIPV anterior(ridge)/posterior/inferior/carina.
The segment of early reconnection | up to 12 months
  Descript as RSPV roof/anterior/posterior/carina, RIPV anterior/posterior/inferior/carina, LSPV roof/anterior(ridge)/posterior/carina, LIPV anterior(ridge)/posterior/inferior/carina.
1-year AF recurrence | up to 12 months
  Using single lead 3-day holter monitoring.
30-day complication associated with procedure | up to 12 months
  Including puncture site hematoma, puncture site pseudoaneurysm, puncture site AV fistula, stroke, TIA, thromboembolism, and others.

CONTACTS AND LOCATIONS:
Overall Officials: Eue-Keun Choi, M.D. Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No